CLINICAL TRIAL: NCT03281824
Title: Open-Label, Dose Increase and Phase I Study of ALT-P7 to Determine Safety, Tolerability, Pharmacokinetics for HER2 Positive Metastatic Breast Cancer Patients Who Have Progressed on Previous Trastuzumab-Based Therapy
Brief Title: Clinical Study of ALT-P7 to Determine Safety, Tolerability and Pharmacokinetics in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alteogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALT-P7
Record Dates: First submitted 2017-09-05; First posted 2017-09-13 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2 Positive Breast Cancer; ALT-P7; Antibody-Drug Conjugate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALT-P7 (Experimental): * 8 groups: 0.3 mg/kg, 0.6 mg/kg, 1.2 mg/kg, 2.4 mg/kg, 3.6 mg/kg, 4.2 mg/kg, 4.5 mg/kg, 4.8 mg/kg,
  * Administration: Day 1 of each 3-week cycle
  Interventions: Biological: ALT-P7 (HM2-MMAE)

INTERVENTIONS:
Biological: ALT-P7 (HM2-MMAE) — Antibody-Drug Conjugate

SUMMARY:
This open-label study assessed the safety, tolerability and pharmacokinetics of ALT-P7(HM2-Drug Conjugate) in patients with HER2-positive metastatic breast cancer who have progressed on previous Trastuzumab-based therapy. Patients received ALT-P7(0.3 mg/kg~5.4 mg/kg, 7 groups) intravenously on Day 1 of each 3-week cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who voluntarily signed the agreement
2. Adult patients ≥ 19 years of age
3. Eastern Cooperative Oncology Group(ECOG) Performance status of 0 or 1
4. Appropriate organism function proven by the following laboratory test results

   * Absolute neutrophil count ≥ 1500 cells/mm³
   * Platelets ≥ 100,000 cells/mm³
   * Hemoglobin ≥ 9.0 g/dL

     * Patients can receive red blood cell transfusions at this level.
   * Creatinine ≤ 1.5 × Upper Limit of Normal(ULN)
   * Aspartate Transaminase(AST) and Alanine Transaminase(ALT) ≤ 2.5 × ULN
   * Alkaline phosphatase ≤ 2.5 × ULN

     * Patients with liver and/or bone metastases: AST and ALT ≤ 5 × ULN, Alkaline phosphatase ≤ 5 × ULN
   * Albumin ≥ 3.0 g/dL, Total bilirubin ≤ 2.0 mg/dL
   * International Normalized Ratio(INR) < 1.5 × ULN(Except when you are on therapeutic anticoagulation therapy)
5. It should be negative in serum pregnancy test in the case of pre-menopausal women and women who were menopausal for less than 12 months
6. In the case of a fertile woman, it should be negative in pregnancy test, and all men and women should use effective contraceptive methods while enrolled in this study. You must also agree to continue the contraception during the trial and up to 6 months after the last dose of the test
7. Those who are expected to understand and observe the clinical trial plan according to the tester's judgment
8. Those who voluntarily agreed to participate in this clinical trial and signed the agreement

Exclusion Criteria:

* Criteria for disease

  1. Previous history of intolerance to Trastuzumab including Grade 3-4 infusion reaction or hypersensitivity
  2. Previous history of permanent discontinuation of Trastuzumab due to the toxicity
  3. A person who has untreated or symptomatic brain metastasis, or brain metastasis requiring radiation, surgery or corticosteroid therapy to control the brain metastases within 4 weeks of the first administration
  4. Current Grade ≥ 2 (according to National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events(CTCAE) v4.03 of peripheral neuropathy
  5. If the toxicity of the previous treatment is not recovered to baseline level or lower than Grade 1 except for hair loss and peripheral neuropathy
  6. Hypercalcemia requiring bisphosphonate therapy (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN) However, it is allowed if bisphosphonate has been used for bone metastasis
  7. A person who has received clinical trial material, chemotherapy, hormone therapy, radiotherapy, immunotherapy or biological therapy within 3 weeks of the first administration. However, it is required a minimum of 2 weeks after surgery if stereotactic radiosurgery is performed
  8. Previous history of exposure to the cumulative dose of anthracycline (Doxorubicin > 360 mg/m², Epirubicin > 600 mg/m²)
* Criteria for cardio pulmonary function

  1. Unstable ventricular arrhythmia requiring treatment
  2. Previous history of symptomatic congestive heart failure (NYHA Class II-IV)
  3. Previous history of myocardial infarction or unstable angina within 6 months
  4. Cardiac troponin I ≥ 0.2 ng/mL
  5. A person who has inadequate left ventricular ejection fraction(LVEF) within 3 weeks of the first administration, LVEF <50% by echocardiography or Multiple-gated Acquisition(MUGA)
  6. A person who has severe dyspnea or pneumonia requiring continuous oxygen therapy
* Common criteria

  1. Pregnant or breastfeeding
  2. A person who has undergone surgical operation or significant traumatic injury within 30 days before registration, or is expected to require surgical operation during the clinical trial
  3. Previous history of malignant tumors other than breast cancer within 5 years prior to screening (patient who can participate: squamous cell and basal cell carcinoma of the skin, intraepithelial cancer of the cervix, thyroid papillary cancer, or if the tester considers that the risk of relapse is minimum(regard as full recovery) and the sponsor agrees with it)
  4. A person who needs chronic corticosteroid therapy (≥ 10 mg/day prednisone or equivalent volume of other anti-inflammatory corticosteroids)
  5. If the result of human immunodeficiency virus (HIV), active hepatitis B or hepatitis C is positive during screening
  6. Patients with uncontrolled concomitant illnesses, including mental illness/social conditions, which may affect compliance with clinical trial procedures

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
DLT test | 21 days after first administration
  Determination of Maximum Tolerated Dose(MTD) and the dose level showing Dose Limiting Toxicity(DLT), or determination of Recommended Phase II Dose(RP2D) as an alternative to MTD establishment

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 4 weeks
  Evaluate adverse events by the Common Terminology Criteria for Adverse Event (CTCAE v4.03) classification, immune-related adverse events(irAEs)
Pharmacokinetics test | up to 4 weeks
  analyze metabolism and discover the fate of a ALT-P7 from administration up to completely eliminated from the body (Group 3(1.2 mg/kg) ~ Group 7(5.4 mg/kg))
Immunogenicity test | up to 4 weeks
  After administration of the drug for clinical trial, the descriptive statistics of the dose group and the measurement point are calculated
Efficacy test | At the end of Cycle 2 (each cycle is 21 days)
  Provide descriptive statistics for each capacity group(the number of subjects, average, standard deviation, median, minimum value, maximum value)

CONTACTS AND LOCATIONS:
Locations (1):
- Alteogen, Daejeon, South Korea